CLINICAL TRIAL: NCT01455363
Title: Etude peropératoire de la Perfusion Sanguine Des Carcinomes Basocellulaires Par Imageur Laser Doppler, au Cours de la Manipulation de l'Influx artériel Tumoral - Recherche d'un phénomène d'hyperémie Tumorale Post-occlusive
Brief Title: Post-occlusive Reactive Hyperemia and Basal-cell Carcinoma
Acronym: HPOB
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut Curie (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: IC 2011-01
Record Dates: First submitted 2011-10-10; First posted 2011-10-19 (Estimated); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Carcinoma, Basal Cell
MeSH Terms: conditions — Carcinoma, Basal Cell | interventions — Laser Speckle Contrast Imaging

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: BCC surgery — This clinical trial will use skin flap model for trunk and facial BCC, with respect the classical excision margin of BCC surgery (3-4mm): after local anesthesia, a little random pattern skin flap will be raised around the BCC, then the cutaneous pedicle will be clamped with surgical clamp for 3 minutes and clamp released.
Other: Tourniquet ischemia — In case of limb BCC, limb tourniquet will be used, and occluded during 3 minutes upstream to the BCC location.
Other: Laser speckle imaging — During all steps of experimentation, laser speckle imaging will be used to measure continuously the peri-tumoral and tumoral perfusion, start from tumor excision, up to10 minutes after tumor pedicle clamp or tourniquet release.

SUMMARY:
The investigators aim to test the hypothesis and to proof thank to laser speckle contrast imaging that post-occlusive reactive hyperemia (PORH) can be induced through a tumor, in this case, through a basal cell carcinoma, which will be used as a model of study of tumor vasculature.

This new concept of tumor perfusion artificial increase could be used in the future for malignant tumors treatment, in order to increase tumor mean oxygen partial pressure (thus decreasing tumor hypoxia, hallmark of malignant tumors) during cancerology therapies, like radiotherapy and/or chemotherapy, and increase their efficacy.

This clinical trial will use skin flap model for trunk and facial basal cell carcinoma (BCC), with respect the classical excision margin of BCC surgery (3-4mm): after local anesthesia, a little random pattern skin flap will be raised around the BCC, then the cutaneous pedicle will be clamped with surgical clamp for 3 minutes and clamp released.

In case of limb BCC, limb tourniquet will be used, and occluded during 3 minutes upstream to the BCC location.

During all steps of experimentation, laser speckle imaging will be used to measure continuously the peri-tumoral and tumoral perfusion, start from tumor excision, up to10 minutes after tumor pedicle clamp or tourniquet release.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18
* Histologically proved cutaneous BCC
* Patient being informed and having signed the consent to participate to the study

Exclusion Criteria:

* Counter-indication to surgery
* Patient being unable to attend future follow-up visits
* Patient with severe cognitive impairment
* Patient not affiliated to a social security regimen
* Patient with limb BCC and history of peripheral vascular artery surgery like bypass and/or vascular prothesis on the same limb (tourniquet counter-indication)
* Local bone invasion of BCC detected with imagery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2011-06; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
Evaluation of blood perfusion of tumor as ROI (Region Of Interest) | 5 months
  Evaluation of blood perfusion of tumor as ROI (Region Of Interest)in unit of laser doppler perfusion, analyzed by the software Pimsoft with the imager laser doppler Pericam PSI system of Perimed.

CONTACTS AND LOCATIONS:
Overall Officials: GUILHARD Thierry, MD, Principal Investigator — INSTITUT CURIE - HOPITAL RENE HUGUENIN
Locations (1):
- Institut Curie, Paris, France

REFERENCES:
- [Result] Reyal J, Lebas N, Fourme E, Guihard T, Vilmer C, Le Masurier P. Post-occlusive reactive hyperemia in basal cell carcinoma and its potential application to improve the efficacy of solid tumor therapies. Tohoku J Exp Med. 2012 Jun;227(2):139-47. doi: 10.1620/tjem.227.139. PMID 22706476